CLINICAL TRIAL: NCT02698046
Title: Oral Iron Therapy in Chronic Heart Failure Patients: a Randomized, Placebo-controlled and Double-blind Clinical Trial (Pilot Study) of Efficiency
Brief Title: Oral Iron Therapy in Chronic Heart Failure Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Jaqueline Rodrigues de Souza Gentil, Master degree, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13/03301-1
Record Dates: First submitted 2015-12-16; First posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure
Keywords: Heart failure; Iron; Anemia; Chronic disease
MeSH Terms: conditions — Heart Failure; Anemia; Chronic Disease | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferrous sulfate (Experimental)
  Interventions: Dietary Supplement: Ferrous sulfate
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo starch

INTERVENTIONS:
Dietary Supplement: Ferrous sulfate — 200mg of ferrous sulfate three times a day for 4 months
  Arms: Ferrous sulfate
Dietary Supplement: Placebo starch — 200mg of placebo starch three times a day for 4 months
  Arms: Placebo

SUMMARY:
This study is design to evaluate the effectiveness of oral iron therapy in patients with heart failure and identify the central and peripheral mechanisms involved in the improvement of functional capacity after intervention. The investigation includes subjective and objective measures on exercise performance and heart function after intervention, and the tolerability of oral iron treatment.

DETAILED DESCRIPTION:
This is a placebo-controlled, double-blind and randomized clinical trial that will include patients with symptomatic stable chronic heart failure (New York Heart Association Functional Class II or III), with diagnosis of iron deficiency (ferritin <100 ng / dL or ferritin between 100 - 300 ng / dL and transferrin saturation <20%) followed in an outpatient clinic. The enrolled patients (n = 36) will be randomly allocated in the ratio 2:1 to treatment with 60 mg of elemental iron orally (n = 24) or placebo administration (n = 12), 3 times daily for 4 months. The primary outcome investigated will be an increase of the transferrin saturation ≥ 10 percentage points between baseline and after the intervention. Secondary outcomes of the study will be the change in iron stores, red blood cell indices, neurohumoral activation, left ventricular systolic function, functional capacity, mechanoreflex activity, and quality life score.

ELIGIBILITY:
Inclusion criteria

* Both gender patients aged over 18 years;
* Diagnosis of chronic heart failure (identified by the use of Framingham criteria) for ≥ 6 months;
* New York Heart Association functional class II and III;
* Left ventricular ejection fraction ≤ 45%
* Regular attendance in an outpatient Heart Failure Clinic;
* Adequate therapeutic drug for heart failure syndrome based on beta-adrenergic blocker, angiotensin converting enzyme inhibitor or angiotensin receptor blocker, and mineralocorticoid receptor blocker;
* Evidence of iron deficiency in biochemical analyses: ferritin values < 100 ng/dL or between 100 ng/dL and 300 ng/dL, with transferrin saturation < 20%;
* Hemoglobin value between 9,0 - 16 g/dL;
* Provide written informed consent.

Exclusion criteria

* Recent device implant (in the last 3 months) or perspective of device implantation (conventional or multisite pacing) in the next 6 months;
* Known active infection, inflammatory disease or C-reactive protein > 20 mg/dL
* Immunosuppressive therapy;
* In use of erythropoietin and/or current treatment with oral or intravenous iron;
* Clinically bleeding or blood transfusion in previous 3 months;
* Renal failure on dialysis;
* Hemoglobinopathies, hemochromatosis or active malignancy;
* Unstable angina pectoris or clinically significant uncorrected valvular disease, except mitral and tricuspid regurgitation secondary to ventricular dilatation;
* Acute myocardial infarction or acute coronary syndrome, transient ischaemic attack within the last 3 months;
* Uncontrolled arterial hypertension;
* Evidence of comorbidity that features active systemic disease, i.e. liver disease, collagen disease and untreated hyperthyroidism or hypothyroidism;
* Pregnant or lactating women;
* Anaemia due to reasons other than iron deﬁciency (i.e. vitamin B12 deficiency);
* Recent admission for decompensated heart failure (last 3 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-06 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Biochemical parameter of serum transferrin saturation | 4 months

SECONDARY OUTCOMES:
Biochemical parameter of hemoglobin in the hemogram analysis | 4 months
Biochemical parameter of serum ferritin | 4 months
Volume of oxygen consumed at peak exercise during cardiopulmonary exercise testing | 4 months
  Unit of measure mL/kg/min
Volume of oxygen consumed at anaerobic threshold during cardiopulmonary exercise testing | 4 months
  Unit of measure mL/kg/min
Ejection fraction of the left ventricle on doppler echocardiographic study | 4 months
  Unit of measure %
Biochemical parameter of N-terminal pro-brain natriuretic peptide (NT-pro-BNP) serum levels | 4 months
Blood pressure results during mechanoreflex evaluation | 4 months
  Unit of measure mmHg
Heart rate results during mechanoreflex evaluation | 4 months
  Unit of measure beats per minute
Volume of oxygen consumed results during mechanoreflex evaluation | 4 months
  Unit of measure mL/kg/min
Total score of physical, emotional, and overall dimensions domains of the Minnesota Living with Heart Failure Questionnaire | 4 months
  Score range 0 to 105 points

OTHER OUTCOMES:
Biochemical parameter of serum urea | 4 months
  Unit of measure mg/dL
Biochemical parameter of serum creatinine | 4 months
  Unit of measure mg/dL
Biochemical parameter of serum sodium | 4 months
  Unit of measure mg/dL
Biochemical parameter of serum potassium | 4 months
  Unit of measure mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Jaqueline RS Gentil, Master, Principal Investigator — University of Sao Paulo
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anker SD, Comin Colet J, Filippatos G, Willenheimer R, Dickstein K, Drexler H, Luscher TF, Bart B, Banasiak W, Niegowska J, Kirwan BA, Mori C, von Eisenhart Rothe B, Pocock SJ, Poole-Wilson PA, Ponikowski P; FAIR-HF Trial Investigators. Ferric carboxymaltose in patients with heart failure and iron deficiency. N Engl J Med. 2009 Dec 17;361(25):2436-48. doi: 10.1056/NEJMoa0908355. Epub 2009 Nov 17. PMID 19920054
- [Background] Jankowska EA, Rozentryt P, Witkowska A, Nowak J, Hartmann O, Ponikowska B, Borodulin-Nadzieja L, Banasiak W, Polonski L, Filippatos G, McMurray JJ, Anker SD, Ponikowski P. Iron deficiency: an ominous sign in patients with systolic chronic heart failure. Eur Heart J. 2010 Aug;31(15):1872-80. doi: 10.1093/eurheartj/ehq158. Epub 2010 Jun 21. PMID 20570952
- [Background] Okonko DO, Mandal AK, Missouris CG, Poole-Wilson PA. Disordered iron homeostasis in chronic heart failure: prevalence, predictors, and relation to anemia, exercise capacity, and survival. J Am Coll Cardiol. 2011 Sep 13;58(12):1241-51. doi: 10.1016/j.jacc.2011.04.040. PMID 21903058